CLINICAL TRIAL: NCT01790490
Title: The Effect of Ketamine on Reducing Cue Reactivity in Cocaine Users
Brief Title: Glutamatergic Modulation of Cocaine-related Deficits
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: #6162
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2016-06-27 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ketamine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- K1 (Experimental): Ketamine 0.41 mg/kg infused over 52 min (K1)
  Interventions: Drug: Ketamine 0.41 mg/kg
- K2 (Experimental): Ketamine 0.71 mg/kg infused over 52 min (K2)
  Interventions: Drug: Ketamine 0.71 mg/kg
- LZP (Experimental): Lorazepam 2 mg infused over 52 minutes (LZP)
  Interventions: Drug: Lorazepam 2 mg

INTERVENTIONS:
Drug: Ketamine 0.41 mg/kg — 52 minute iv infusion of ketamine 0.41 mg/kg
  Other Names: K1
  Arms: K1
Drug: Ketamine 0.71 mg/kg — 52 minute iv infusion of ketamine 0.71 mg/kg. This dose follows K1 in all 3 orderings.
  Other Names: K2
  Arms: K2
Drug: Lorazepam 2 mg — 52 minute infusion of lorazepam 2 mg. This serves as an active control.
  Other Names: LZP
  Arms: LZP

SUMMARY:
Cocaine dependence involves problematic neuroadaptations, such as heightened reactivity to cocaine cues, that may be responsive to pharmacological modulation of glutamatergic circuits. Despite promising preclinical findings with n-methyl-d-aspartate receptor (NMDAr) modulators, studies with human subjects have been unsuccessful to date. The purpose of this investigation is to examine the effects of the NMDAr antagonist ketamine, recently found to have potent therapeutic effects in humans, on cue-induced craving and impaired motivation for quitting cocaine in cocaine dependent participants, 24-hours post-infusion.

DETAILED DESCRIPTION:
In this study, volunteers will undergo a 9 day inpatient trial during which they will receive three counter-balanced infusions (two doses of ketamine and a dose of lorazepam) on three separate days in a within-subject, double-blind, controlled design. Of the various glutamate antagonists available for human use, ketamine will be utilized because its safety profile, pharmacokinetics, and range of tolerable sub-anesthetic dosings have been very well studied. Also, ketamine has shown promise in managing opiate and alcohol use disorders in certain studies, and may therefore be the most likely glutamate antagonist to dampen cue reactivity and increase motivation in cocaine users. If ketamine significantly improves these deficits, this would suggest that the drug should be investigated further for potential utility as a treatment for cocaine dependence.

ELIGIBILITY:
Inclusion Criteria

1. Active free-base cocaine dependence (at least 4 days of use over the past month, with at least 1 use per week); if the participant uses through another route (IN, IV), then the FB route is dominant (> 80% of occasions).
2. Physically healthy
3. No adverse reactions to study medications
4. 21-52 years of age
5. Normal body weight
6. Responsive to drug cues
7. Capacity to consent

Exclusion Criteria:

1. Seeking treatment or abstinence
2. DSM IV criteria for substance dependence (other than methamphetamine, cocaine, cannabis, or nicotine), or DSM IV criteria for abuse of ketamine or lorazepam
3. DSM-IV criteria for other Axis I psychiatric illness that may make participation hazardous such as schizophrenia, schizoaffective disorder, psychosis NOS, MDD, psychosis secondary to substances, or bipolar disorder
4. Delirium, Dementia, Amnesia, Cognitive Disorders, or dissociative disorders
5. Current suicide risk or a history of suicide attempt within the past 2 years
6. Current use of prescribed psychotropic medication
7. Pregnancy, nursing, or had a baby within the past 6 mo.
8. Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
9. Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), anemia, active hepatitis or other liver disease, or diabetes
10. "Bad" reaction/experience with prior exposure to ketamine or lorazepam
11. History of significant violence
12. First degree relative with a psychotic disorder

Ages: 21 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI/Columbia College of Physicians and Surgeons; Carl Hart, PhD, Study Chair — NYSPI/Columbia College of Physicians and Surgeons
Locations (1):
- NYSPI, New York, New York, United States

REFERENCES:
- [Derived] Dakwar E, Levin F, Foltin RW, Nunes EV, Hart CL. The effects of subanesthetic ketamine infusions on motivation to quit and cue-induced craving in cocaine-dependent research volunteers. Biol Psychiatry. 2014 Jul 1;76(1):40-6. doi: 10.1016/j.biopsych.2013.08.009. Epub 2013 Sep 12. PMID 24035344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using advertisements and were seen at NYSPI.
Pre-assignment Details: Participants were excluded if they could not comply with study procedures or if they were found to be ineligible.
Groups:
- K1, LZP, and K2: Ketamine 0.41 (K1) followed by lorazepam (LZP) and then ketamine 0.71. Infusions are separated by 48 hours. This ordering allows for comparison between K1 and LZP, and between the post-K1 additive effects of LZP and K2.
- LZP, K1, and K2: LZP followed by K1 and then K2. Infusions are separated by 48 hours. This order allows for comparison between LZP and K1.
- K1, K2, and LZP: K1 followed by K2 and then LZP. Infusions are separated by 48 hours. This allows for within-subject comparison of the post-K1 additive effects of K2 and LZP.
Period: Overall Study
Arm/Group | K1, LZP, and K2 | LZP, K1, and K2 | K1, K2, and LZP
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | K1, LZP, and K2 | LZP, K1, and K2 | K1, K2, and LZP | Total
Number analyzed (Participants) | 3 | 3 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9) | 48.2 (6.1) | 44.2 (8.2) | 47.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 2 | 3 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Cue Reactivity
Description: Serial visual analogue scale (VAS) scores for craving elicited by cocaine cue: units on a scale (0-200), high is worse. Scores are obtained at baseline and at 24 hours after the infusion.
Time Frame: Baseline and 24 hours after infusion
Measure: Median (Standard Error); unit: units on a scale (0-200), high is worse
Groups:
- Ketamine Infusion 0.41 mg/kg Over 52 Minutes (K1): Ketamine 0.41 mg/kg infused over 52 min (K1)
  Ketamine 0.41 mg/kg: 52 minute iv infusion of ketamine 0.41 mg/kg
- Ketamine Infusion 0.71 mg/kg Over 52 Minutes (K2): Ketamine 0.71 mg/kg infused over 52 min (K2)
  Ketamine 0.71 mg/kg: 52 minute iv infusion of ketamine 0.71 mg/kg. This dose follows K1 in all 3 orderings.
- Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP): Lorazepam 2 mg infused over 52 minutes (LZP)
  Lorazepam 2 mg: 52 minute infusion of lorazepam 2 mg. This serves as an active control.
Arm/Group | Ketamine Infusion 0.41 mg/kg Over 52 Minutes (K1) | Ketamine Infusion 0.71 mg/kg Over 52 Minutes (K2) | Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP)
Number analyzed (Participants) | 8 | 8 | 8
units on a scale (0-200), high is worse | 126 (66) | 18 (13) | 16 (12)

2. Primary Outcome: Change in Motivation to Quit
Description: Motivation score obtained from the University of Rhode Island Change Assessment (URICA). Scores are obtained at baseline and at 24 hours after each infusion. The scores are 0-13, with higher scores indicating greater motivation. The analysis is within-subject. Scores included below are means; higher scores represent higher motivation to quit than do lower scores.
Time Frame: Baseline and 24 hours post-infusion
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Ketamine Infusion 0.41 mg/kg Over 52 Minutes (K1): Ketamine 0.41 (K1) followed by lorazepam (LZP) and then ketamine 0.71. Infusions are separated by 48 hours. This ordering allows for comparison between K1 and LZP, and between the post-K1 additive effects of LZP and K2.
- Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP): LZP followed by K1 and then K2. Infusions are separated by 48 hours. This order allows for comparison between LZP and K1.
- Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP) Following K1: Infusions are separated by 48 hours. This allows for within-subject comparison of the post-K1 additive effects of K2 and LZP.
Arm/Group | Ketamine Infusion 0.41 mg/kg Over 52 Minutes (K1) | Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP) | Lorazepam Infusion 2 mg/kg Over 52 Minutes (LZP) Following K1
Number analyzed (Participants) | 3 | 3 | 2
units on a scale | 4.35 [2.12 to 6.01] | 3.2 [1.1 to 5.87] | 4.2 [2.12 to 6.56]

ADVERSE EVENTS:
Groups:
- Ketamine 0.41 (K1): Ketamine 0.41 (K1) over 52 minutes
- Lorazepam 2 mg (LZP): Lorazepam 2 mg (LZP) over 52 minutes
- Ketamine 0.71 (K2): Ketamine 0.71 mg/kg over 52 minutes (K2)
Arm/Group | Ketamine 0.41 (K1) | Lorazepam 2 mg (LZP) | Ketamine 0.71 (K2)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No